CLINICAL TRIAL: NCT02564107
Title: An Open Label Study of the Efficacy, Safety, and Pharmacoeconomics of Oral Ibandronate (Bondronat 50 mg) in Treatment of Metastatic Bone Disease
Brief Title: A Study of Ibandronate (Bondronat) in Participants With Metastatic Bone Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18044
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Pain; Bone Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Pain; Bone Neoplasms; Neoplasm Metastasis | interventions — Ibandronic Acid

ARMS (1):
- Ibandronate (Experimental): Female participants with metastatic bone disease secondary to breast cancer will receive ibandronate for a period of 25 weeks.
  Interventions: Drug: Ibandronate

INTERVENTIONS:
Drug: Ibandronate — Participants will receive ibandronate, 50 milligrams (mg) by mouth every morning, for a period of 25 weeks.
  Other Names: Bondronat

SUMMARY:
This study will evaluate the efficacy, safety, and effect on quality of life of oral ibandronate (Bondronat) in participants with breast cancer and metastatic bone disease. The anticipated time on study treatment is 25 weeks, and the target sample size is 50 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Females at least 18 years of age
* Breast cancer
* Bone metastases

Exclusion Criteria:

* Use of bisphosphonates within the last 3 months
* Prior use of gallium nitrate or metastron
* Severely impaired renal function
* Hypocalcemia or primary hyperparathyroidism
* Central nervous system (CNS) metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-11; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of skeletal events according to Skeletal Morbidity Period Rate (SMPR) | Up to 25 weeks

SECONDARY OUTCOMES:
Incidence of bone pain according to participant questionnaire | Up to 25 weeks
Analgesic consumption according to participant questionnaire | Up to 25 weeks
Change in serum pyridinoline cross-linked carboxyterminal telopeptide of collagen type I (ICTP) | Up to 25 weeks
Short Form 36 (SF-36) score | Up to 25 weeks
Incidence of adverse events (AEs) | Up to approximately 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (6):
- Bulgaria (6):
  - Plovdiv
  - Shumen
  - Sofia
  - Stara Zagora
  - Varna
  - Veliko Tarnovo